CLINICAL TRIAL: NCT03577184
Title: Effect of Vildagliptin & Metformin Combination on Glycemic Control and Hypoglycemic Episodes. An Observational Real Life Trial
Brief Title: Evaluating the Glycemic Control wIth Vildagliptin and Metformin Combination Therapy.
Acronym: GRIP
Status: Withdrawn | Type: Observational
Why Stopped: Institutions issue
Sponsor: Clinision (Other)
Responsible Party: Sponsor
Other Study IDs: CN/PK/GRIP/SP/2017-01
Record Dates: First submitted 2018-01-18; First posted 2018-07-05 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GRIP, DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Vildagliptin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Metformin/Vildagliptin — Vildagliptin belongs to dipeptidyl peptidase-4 (DPP-4) inhibitor. Inhibition of dipeptidyl peptidase-4 (DPP-4) and metformin is a Biguanides.
  Other Names: Galvecta Plus

SUMMARY:
To evaluate the changes from baseline in random blood sugar (RBS) and fasting blood sugar (FBS) levels at week 12 in participants receiving Vildagliptin combination with Metformin.

DETAILED DESCRIPTION:
Galvecta Plus is a combination of Vildagliptin and Metformin hydrochloride. Combination drug with complementary mechanisms of action, provides efficacy and allows to reach glycemic targets compared to continuing metformin monotherapy and is used as an oral hypoglycemic in Type II diabetes mellitus that shows potential to achieve better blood glucose without increasing the risk of hypoglycemia, exposing to weight gain and altering common cardiovascular risk factors (hypertension and lipid profile). The fact that Vildagliptin with metformin substantially enhances the incretin effect. Vildagliptin belongs to dipeptidyl peptidase-4 (DPP-4) inhibitor. Inhibition of dipeptidyl peptidase-4 (DPP-4) by Vildagliptin prevents degradation of glucagon-like peptide-1 (GLP-1) and reduces glycaemia in patients with type 2 diabetes mellitus, with low risk for hypoglycemia and no weight gain and metformin is a Biguanides with antihyperglycaemic effects, lowering both basal and postprandial plasma glucose. It does not stimulate insulin secretion and therefore does not produce hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with type 2 diabetes mellitus (DM).
* Patient with HbA1c levels greater than 7.0% who were naïve or were receiving monotherapy with oral hypoglycemic agent were eligible to participate in the study.

Exclusion Criteria:

* Patient with a history diabetic ketoacidosis, clinically significant liver or renal disease, congestive heart failure requiring pharmacological treatment, coronary artery percutaneous intervention or unstable angina within the past 6 month excluded from study
* Participants who are pregnant or with gestational DM
* Age over 80 years
* Hypersensitivity to any active ingredient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes Mellitus patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Random blood sugar (RBS) and fasting blood sugar (FBS) levels at week 12 in participants receiving Vildagliptin combination with Metformin | Week 12
  To determine the efficacy of vildagliptin/metformin changes from baseline in random blood sugar (RBS) and fasting blood sugar (FBS) levels after 12 weeks of therapy.
  [Designated as safety issue: No ]

SECONDARY OUTCOMES:
Changes from baseline in HbA1c Levels at Week 12 in participants receiving Vildagliptin combination with Metformin | Week 12
  To determine the efficacy of vildagliptin/metformin changes from baseline in HbA1c levels after 12 weeks of therapy.
  [ Designated as safety issue: No ]
Number of participants experiencing hypoglycemic episodes in the 12 weeks receiving Vildagliptin combination with Metformin. | Week 12
  To evaluate the number of participants experiencing hypoglycemic episodes in the 12 weeks [ Designated as safety issue: Yes ]
Number of participants who experienced an Adverse Event | 12 weeks
  To evaluate the number of participants who experienced an adverse event after 12 weeks of therapy.
  [ Designated as safety issue: Yes ]